CLINICAL TRIAL: NCT00448305
Title: An Open-label, Randomized, Controlled Phase-II Trial Evaluating the Efficacy and Safety of EndoTAG-1 in Triple Receptor Negative Breast Cancer Patients
Brief Title: EndoTAG-1 in Triple Receptor Negative Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT 4002; EudraCT-Nr. 2006-002221-23
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; metastatic; relapsed; triple-receptor negative; EndoTAG-1; metastatic or relapsed breast neoplasm
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Recurrence | interventions — MBT-0206; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): EndoTAG-1 + Paclitaxel
  Interventions: Drug: EndoTAG-1 + paclitaxel
- 2 (Experimental): EndoTAG-1
  Interventions: Drug: EndoTAG-1
- 3 (Active Comparator): Paclitaxel
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: EndoTAG-1 + paclitaxel — EndoTAG-1 22 mg/m² + Paclitaxel 70 mg/m² weekly
  Arms: 1
Drug: EndoTAG-1 — EndoTAG-1 44 mg/m² twice weekly
  Arms: 2
Drug: Paclitaxel — Paclitaxel 90 mg/m² weekly
  Arms: 3

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of a therapy with EndoTAG-1 + paclitaxel in combination and EndoTAG-1 alone as a rescue therapy for patients with relapsed or metastatic triple receptor negative breast cancer (a special subgroup of breast cancer).

DETAILED DESCRIPTION:
Breast cancer is still a major public health problem worldwide, as it is by far the most frequent neoplasm in women. In recent years so-called "profiling of breast cancer" with expression arrays has become common and it was suggested that the results will allow individualization of care. Breast cancer may now be subclassified into luminal, basal, and HER-2 subtypes with distinct differences in prognosis and response to therapy. About 80% of all basal-like-breast cancers possess a so-called "triple-receptor-negative" phenotype.

Patients with "triple receptor negative breast cancer" have a complete absence of hormone receptors incl. HER-2, an aggressive clinical course and a paucity of treatment options. The only therapeutic option is chemotherapy and in this respect the choice of cytostatic agents is limited. Against this background, the study tries to find another therapeutic option by combining a vascular-disrupting activity with the cytostatic effects of paclitaxel in the study drug EndoTAG-1.

Comparison: EndoTAG-1 + paclitaxel (combination therapy) and EndoTAG-1 (monotherapy) in comparison to paclitaxel (control group)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven triple-receptor-negative metastatic or relapsed breast cancer
* Minimum interval of 6 months after the end of any previous taxane- containing chemotherapy regimen
* At least one tumor lesion measurable according to RECIST criteria
* Gender: female
* Age >= 18 years old
* Negative pregnancy test (females of childbearing potential)
* Willingness to perform double-barrier-contraception during study and for 6 months post chemotherapy treatment
* ECOG performance status 0, 1 or 2
* Signed informed consent

Exclusion Criteria:

* More than 1 previous chemotherapeutic treatment for metastatic or relapsed disease
* Major surgery < 4 weeks prior to enrollment
* Immunotherapy < 2 weeks prior to enrollment
* Severe pulmonary obstructive or restrictive disease
* Uncontrolled inflammatory disease (autoimmune or infectious)
* Clinically significant cardiac disease (NYHA stadium > 2)
* Laboratory tests (hematology, chemistry) outside specified limits
* Pregnancy or nursing status
* Known positive HIV testing
* Known hypersensitivity to any component of the EndoTAG-1 or taxane formulations
* History of malignancy other than breast cancer < 5 years prior to enrollment, except skin cancer (i.e. basal or squamous cell carcinoma) treated locally
* Known progressive cerebral metastasis (patients with cerebral metastases in a stable state or after successful surgical or radiological treatment are allowed to participate in the study)
* History of active or significant neurological disorder or psychiatric disorder that would prohibit the understanding and giving of informed consent, or would interfere in the clinical and radiological evaluation of central nervous system during the trial
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
4-month progression free survival (PFS) rate | 4 month

SECONDARY OUTCOMES:
median progression free survival (PFS) time | progression of last patient
tumor response | Last patient out
4-month survival rate | 4-month
median overall survival time | Withdrawal or death of last patient
pain assessment | Last patient out
clinical benefit assessment via quality of life (QoL)Scale | Last patient out
adverse events | Last patient out
laboratory values | Last patient out
dose variations | Last patient out

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Awada, Dr., Principal Investigator — Institut Jules Bordet - Centre des Tumeurs de l'Université Libre de Bruxelles, 121 Boulevard de Waterloo, 1000 Brussels, Belgium
Locations (33):
- Belgium (4):
  - Institut Jules Bordet - Centre des Tumeurs de l'Université Libre de Bruxelles, Brussels
  - CHU Brugmann, Brussels
  - UZ Antwerpen, Edegem
  - CHU Liège, Liège
- France (5):
  - Centre Oscar Lambret, Lille
  - Cente Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hôpital de Jour Centre Henri Kaplan, Tours
  - Institut Gustave Roussy, Villejuif
- India (6):
  - Vedanta Institute of Medical Science, Ahmedabad
  - Bangalore Institute of Oncology, Bangalore
  - Searoc Cancer Center, Jaipur
  - Lakeshore Hospital, Kochi
  - Deenanath Mangeshkar Hospital, Pune
  - Kaushalya Medical Foundation, Thane
- Poland (5):
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Gliwice
  - Instytut im. M. Sklodowskiej-Curie, Lublin
  - NZOZ Grupowa Specjalistyczna, Olsztyn
  - Klinika Onkologii Adadmii Medycznej, Poznan
- Romania (5):
  - Institute of Oncology "Prof. Dr. Al. Trestioreanu", Bucharest
  - Institute of Oncology "Prof. Dr. I. Chiricuta", Cluj-Napoca
  - Center of Medical Oncology, Iași
  - Emergency County Hospital Sibiu, Sibiu
  - Oncology Clinic "Oncomed", Timișoara
- Ukraine (8):
  - Dnepropetrovsk State Medical Acedamy, Dnipro
  - Institute of Medical Radiology of Acedamy of Medical Sciences, Kharkiv
  - Department of Abdominal Surgery, Kiev
  - Institut of Oncology, Kiev
  - Surgical Department, Kiev
  - Rivne Regional Oncological Dispensary, Rivne
  - Sumy Reginal Oncology Center, Sumy
  - Regional Clinical Oncological Dispensary, Uzhhorod

REFERENCES:
- [Derived] Awada A, Bondarenko IN, Bonneterre J, Nowara E, Ferrero JM, Bakshi AV, Wilke C, Piccart M; CT4002 study group. A randomized controlled phase II trial of a novel composition of paclitaxel embedded into neutral and cationic lipids targeting tumor endothelial cells in advanced triple-negative breast cancer (TNBC). Ann Oncol. 2014 Apr;25(4):824-831. doi: 10.1093/annonc/mdu025. PMID 24667715